CLINICAL TRIAL: NCT00306293
Title: The Effect of Valacyclovir 1g Once Daily on HSV-2 Viral Shedding in Subjects Newly Diagnosed With Genital Herpes Infection
Brief Title: VALTREX(Valacyclovir) Once Daily for Viral Shedding In Subjects Newly Diagnosed With HSV-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VLX105832
Record Dates: First submitted 2006-03-21; First posted 2006-03-23 (Estimated); Results first posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2017-08

CONDITIONS: Herpes Labialis
Keywords: Recurrent Genital Herpes
MeSH Terms: conditions — Herpes Labialis; Herpes Genitalis | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: valacyclovir — valacyclovir

SUMMARY:
Eligible subjects will be randomized to receive VALTREX 1g or placebo once daily for 60 days in a two-way crossover study with a washout period of 7 days in between.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in overall general good health.
* If female, subject must be of:

  1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal or surgically sterile); or
  2. Childbearing potential, but must have a negative pregnancy test at randomization, and must be compliant with one of the following: Complete abstinence from intercourse for two weeks before exposure to the study drug, throughout the clinical trial, and for a period of 1 week after study completion or premature discontinuation from the study (to account for elimination of the drug); Have a male partner who is confirmed to be sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject; Use of contraceptive(s) with a documented failure rate of less than 1% per year, including but not limited to: implants of levonorgestrel, use of injectable progestogen, oral contraceptives (either combined or progestogen only), an intrauterine device (IUD) or spermicide plus a mechanical barrier (condom/diaphragm).
* Subjects must be newly diagnosed with a first recognized episode of genital herpes as described in (a) or (b) below (See Appendix 3): a.HSV-2 seropositive at screen, with documented clinical signs and symptoms consistent with genital herpes at screen or within 4 months prior to randomization or b.HSV-2 seronegative at screen, AND HSV-2 culture positive or HSV-2 PCR positive with documented clinical signs and symptoms consistent with genital herpes at screen or within 4 months prior to randomization.
* Subject must be willing and able to provide written informed consent and comply with the protocol.

Exclusion Criteria:

* Subject is known or suspected to be immunocompromised (e.g., subjects receiving immunosuppressive therapy or chemotherapy for malignancy, or are seropositive for HIV).
* Subject received an investigational drug in the 30 days prior to the randomization visit.
* Subject is receiving systemic antiviral or immunomodulatory treatments.
* Subjects who have received systemic antiherpetic treatments (e.g., valacyclovir, acyclovir, ganciclovir, famciclovir) within 3 days of starting study drug, or immunomodulatory treatments in the 30 days before starting study drug.
* Subject has clinically significantly impaired renal function as defined by creatinine clearance less than 50ml/min (calculated using the Cockcroft-Gault formula).
* Subjects with a history or evidence of decompensated liver disease, or clinically significantly impaired hepatic function defined as an ALT (alanine transaminase) level >3 times the normal upper limit.
* Subject is known to be hypersensitive to valacyclovir, acyclovir, ganciclovir or famciclovir.
* Subject has malabsorption or vomiting syndrome or other gastrointestinal dysfunction that may impair drug pharmacokinetics.
* Female subject who is contemplating pregnancy within the duration of the study drug dosing period.
* Female subject who is pregnant and/or nursing.
* Subject with current alcohol or drug abuse.
* Subjects who have received suppressive (daily) therapy for genital herpes prior to randomization. Suppressive therapy is defined as daily antiherpetic therapy of at least 4 weeks duration.
* Subjects with a history of ocular HSV (herpes simplex virus) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-02-20 (Actual); Primary Completion 2006-11-27 (Actual); Study Completion 2006-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- United States (17):
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Carmichael, California
  - GSK Investigational Site, Fair Oaks, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Portage, Michigan
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: VLX105832 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: VLX105832 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: VLX105832 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: VLX105832 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: VLX105832 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: VLX105832 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: VLX105832 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seventy participants were enrolled at 14 centers in the United States. The study was conducted between 20 February 2006 and 28 November 2006.
Pre-assignment Details: Out of the 70 participants 35 participants were randomized to the VALTREX 1 g First then Placebo treatment sequence (VAL-PBO) and 35 participants were randomized to the Placebo first then VALTREX 1 g treatment sequence (PBO-VAL).
Groups:
- VALTREX 1 g First Then Placebo: Participants received VALTREX 1 g (2 x500 mg caplets), OD, orally, for 60 days in first period followed by matching placebo 2 caplets, OD, orally, for 60 days in period second period. The two treatment periods were separated by washout period of seven days.
- Placebo First Then VALTREX 1 g: Participants received matching placebo 2 caplets, OD, orally, for 60 days in first period followed by VALTREX 1 g (2 x500 mg caplets), OD, orally, for 60 days in second period. The two treatment periods were separated by washout period of seven days.
Period: Period 1 (Day 1 to Day 60)
Arm/Group | VALTREX 1 g First Then Placebo | Placebo First Then VALTREX 1 g
Started | 35 | 35
Completed | 27 | 27
Not Completed | 8 | 8
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 3 | 4
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Positive pregnancy Test | 2 | 2
Period: Washout (Day 61 to Day 66)
Arm/Group | VALTREX 1 g First Then Placebo | Placebo First Then VALTREX 1 g
Started | 27 | 27
Completed | 27 | 27
Not Completed | 0 | 0
Period: Period 2 (Day 67 to Day 126 )
Arm/Group | VALTREX 1 g First Then Placebo | Placebo First Then VALTREX 1 g
Started | 27 | 27
Completed | 24 | 26
Not Completed | 3 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Participant determined HSV-2 negative | 0 | 1
Not completed — Pregnancy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Participants received VALTREX 1 g (2 x500 mg caplets) and matching placebo 2 caplets, orally, OD, for 60 days in a two-way crossover design either in sequence VAL-PBO or PBO-VAL. The two treatment periods were separated by washout period of seven days.
Arm/Group | Overall Study
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: Year] | 30.9 (9.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 28
  American Indian or Alaska Native | 2
  Asian - East Asian Heritage | 2
  White - Arabic/North African Heritage | 1
  White - White/Caucasian/European Heritage | 36
  Mixed Race | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Days of Total Shedding (Clinical and Subclinical) as Determined by Type-specific Polymerase Chain Reaction (PCR) Assay for Herpes Simplex Virus Type 2 (HSV-2)
Description: Each participant's study day were classified as either 'shedding' (positive HSV-2 result), 'no shedding' (negative HSV-2 result), or 'unknown' (swabbing not done or assay result not available) confirmed by PCR. If either the daily genital swab or a lesion swab are positive, the day was classified as 'shedding'. Study shedding day was classified as either 'clinical' (investigator-confirmed presence of genital lesions) or 'subclinical' (no genital lesions) by the investigator during recurrence visits. Percent of days with HSV-2 shedding was defined for each participant as the percent of days with PCR data for which HSV-2 shedding was detected by a positive PCR result, i.e., the number of days with HSV-2 PCR shedding divided by total number of days with PCR data, multiplied by 100. Sum of the percent clinical and nonclinical shedding days was reported as total shedding. Mean percent of days with HSV-2 shedding was reported for each treatment group.
Time Frame: Up to 60 days in each treatment period (Up to 148 days)
Population: Intent to Treat Crossover population comprised of all participants in the Intent to Treat population who had at least one PCR swabbing result in each Treatment Period. Intent to Treat population comprised of all participants who received at least one dose of investigational product.
Measure: Mean (Standard Deviation); unit: Percent of days
Groups:
- VALTREX 1 g, OD: Participants received VALTREX 1 g (2 x500 mg caplets), OD, orally, for 60 days in a two-way crossover design either in sequence VAL-PBO or PBO-VAL. The two treatment periods were separated by washout period of seven days.
- Placebo: Participants received matching placebo 2 caplets, OD, orally, for 60 days in a two-way crossover design either in sequence VAL-PBO or PBO-VAL. The two treatment periods were separated by washout period of seven days.
Arm/Group | VALTREX 1 g, OD | Placebo
Number analyzed (Participants) | 52 | 52
Percent of days | 2.9 (5.6) | 13.5 (16.9)

2. Secondary Outcome: Mean Percent Days Subclinical Shedding (no Genital Lesions Present)
Description: The percent of days with subclinical HSV-2 shedding was defined as the percent of all days with PCR data for which subclinical HSV-2 shedding was detected (shedding in the absence of a genital lesion). Mean percent of days with subclinical HSV-2 shedding was reported for each treatment group. Each participant's study day was classified as either 'shedding' (positive HSV-2 result), 'no shedding' (negative HSV-2 result), or 'unknown' (swabbing not done or assay result not available) confirmed by PCR. If either the daily genital swab or a lesion swab was positive, the day was classified as 'shedding'. Study shedding day was classified as either 'clinical' (investigator-confirmed presence of genital lesions) or 'subclinical' (no genital lesions) by the investigator during recurrence visits.
Time Frame: Up to 60 days in each treatment period (Up to 148 days)
Population: Intent-to-Treat Crossover
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | VALTREX 1 g, OD | Placebo
Number analyzed (Participants) | 52 | 52
Percentage of days | 2.4 (4.8) | 11 (15.1)
Statistical Analysis 1: Comparison: VALTREX 1 g, OD vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test; Percent change from Placebo = -78 — Percent change in days with Subclinical HSV-2 Viral Shedding after VALTREX 1g treatment from the placebo

3. Secondary Outcome: Mean Percent Days Clinical Shedding (Presence of Genital Lesions)
Description: The percent of days with clinical HSV-2 shedding was defined as the percent of all days with PCR data for which clinical HSV-2 shedding was detected (shedding in the presence of a genital lesion). Each participant's study day was classified as either 'shedding' (positive HSV-2 result), 'no shedding' (negative HSV-2 result), or 'unknown' (swabbing not done or assay result not available) confirmed by PCR. If either the daily genital swab or a lesion swab was positive, the day was classified as 'shedding'. Study shedding day was classified as either 'clinical' (investigator-confirmed presence of genital lesions) or 'subclinical' (no genital lesions) by the investigator during recurrence visits. Mean percent of days with clinical HSV-2 shedding was reported for each treatment group.
Time Frame: Up to 60 days in each treatment period (Up to 148 days)
Population: Intent-to-Treat Crossover
Measure: Mean (Standard Deviation); unit: Percentage of Days
Arm/Group | VALTREX 1 g, OD | Placebo
Number analyzed (Participants) | 52 | 52
Percentage of Days | 0.6 (1.7) | 2.4 (4.4)
Statistical Analysis 1: Comparison: VALTREX 1 g, OD vs Placebo; Test type: Superiority or Other; p = 0.014, Wilcoxon Rank Sum; Percent change from Baseline = -77 — Percent change in 'percentage of days with clinical HSV-2 viral shedding', after VALTREX 1g treatment from the placebo

4. Secondary Outcome: Percentage of Participants With no Shedding
Description: The proportion of participants with no shedding was defined as the number of participants with no HSV-2 shedding detected by PCR divided by the total number of participants with PCR data in the Treatment Period. Each participant's study day was classified as either 'shedding' (positive HSV-2 result), 'no shedding' (negative HSV-2 result), or 'unknown' (swabbing not done or assay result not available) confirmed by PCR. If either the daily genital swab or a lesion swab was positive, the day was classified as 'shedding'. Study shedding day was classified as either 'clinical' (investigator-confirmed presence of genital lesions) or 'subclinical' (no genital lesions) by the investigator during recurrence visits. Mean percent of days with no shedding was reported for each treatment group.
Time Frame: Up to 60 days in each treatment period (Up to 148 days)
Population: Intent-to-Treat Crossover
Measure: Number; unit: Percentage of participants
Arm/Group | VALTREX 1 g, OD | Placebo
Number analyzed (Participants) | 52 | 52
Percentage of participants | 60 | 29

5. Secondary Outcome: Percentage of Participants With at Least One Genital Herpes Recurrence
Description: The proportion of participants with at least one genital herpes recurrence was defined as the number of participants with at least one investigator-confirmed genital herpes recurrence divided by the total number of participants with at least one clinic visit in the treatment period.
Time Frame: Up to 60 days in each treatment period (Up to 148 days)
Population: Intent-to-Treat Crossover
Measure: Number; unit: Percetage of participants
Arm/Group | VALTREX 1 g, OD | Placebo
Number analyzed (Participants) | 52 | 52
Percetage of participants | 21 | 48

6. Secondary Outcome: Median Time to First Genital Herpes Recurrence (Days)
Description: Time to first genital herpes recurrence was evaluated using Kaplan-Meier estimates of investigator-confirmed genital herpes recurrences censoring the data from participants who prematurely discontinue the study at the time of discontinuation.
Time Frame: Up to Day 68
Population: First Period Efficacy Population included participants in the Intent to Treat Exposed Population and was used for efficacy analyses restricted to the First Treatment Period.
Measure: Median (Full Range); unit: Days
Arm/Group | VALTREX 1 g First Then Placebo | Placebo First Then VALTREX 1 g
Number analyzed (Participants) | 33 | 35
Days | NA [11 to NA] — Genital herpes did not recur in more than half of participants within the first treatment period. The analysis was restricted to Treatment Period I (60 days) + 7 days of Washout Period. Therefore the median and upper limit could not be estimated. | 61 [4 to 61]

7. Secondary Outcome: Number of Participants With Any Adverse Event (AE) and Serious Adverse Event (SAE)
Description: AE was defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE include adverse events that result in death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. No SAEs were reported in this study.
Time Frame: Up to 148 days
Population: Intent to treat exposed population comprised of all participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | VALTREX 1 g, OD | Placebo
Number analyzed (Participants) | 62 | 62
Participants
  Any AE | 19 | 26
  Any SAE | 0 | 0

ADVERSE EVENTS:
Time Frame: AE and SAE were collected from randomization visit (Day 1) until the recurrence visit (Day 148)
Description: Intent-to-Treat Exposed population was used to collect the AEs and SAEs.
Arm/Group | VALTREX 1 g, OD | Placebo
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62
Other Adverse Events (participants affected / at risk) | 19/62 | 26/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VALTREX 1 g, OD (N=62) | Placebo (N=62)
Fungal infection (Infections and infestations) | 3 | 6
Upper respiratory tract infection (Infections and infestations) | 3 | 1
Sinusitis (Infections and infestations) | 2 | 1
Vaginitis bacterial (Infections and infestations) | 2 | 1
Bronchitis (Infections and infestations) | 2 | 0
Ear infection (Infections and infestations) | 2 | 0
Folliculitis (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 2 | 0
Vulvovaginitis trichomonal (Infections and infestations) | 0 | 2
Anogenital warts (Infections and infestations) | 0 | 1
Cervicitis human papilloma virus (Infections and infestations) | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1
Labyrinthitis (Infections and infestations) | 1 | 0
Onychomycosis (Infections and infestations) | 1 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 1
Sialoadenitis (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 2
Migraine (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Smear cervix abnormal (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 2
Sleep disorder (Psychiatric disorders) | 0 | 1
Stress (Psychiatric disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.